CLINICAL TRIAL: NCT06770660
Title: Evaluating the Effectiveness of Telemedicine-based Exercise Programme in Improving Cardiorespiratory Fitness in Asian Paediatric Population: a Randomised Controlled Trial
Brief Title: Effect of Tele-exercise on Cardiorespiratory Fitness in Paediatrics
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: KK Women's and Children's Hospital (Other Government)
Responsible Party: Principal Investigator, Benny Loo Kai Guo, Senior Consultant, KK Women's and Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 02/FY2024/P2/18-A140
Record Dates: First submitted 2025-01-07; First posted 2025-01-13 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-01

CONDITIONS: Cardiorespiratory Fitness; Insulin Resistance
Keywords: paediatric; cardiorespiratory fitness; telemedicine; insulin resistance
MeSH Terms: conditions — Insulin Resistance | interventions — Telemedicine

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Telemedicine (Experimental): Participants who receive 10-week telemedicine-based exercise programme and physical activity education.
  Interventions: Behavioral: Telemedicine
- Lifestyle (Placebo Comparator): Participants who receive physical activity education only.
  Interventions: Behavioral: Lifestyle

INTERVENTIONS:
Behavioral: Telemedicine — A 10-week telemedicine-based exercise programme consisting of 90-minute sessions conducted weekly via a video conferencing platform.
  All participants will also be educated on physical activity recommendations, including achieving a minimum of 12,000 steps daily, and required to perform weekly check-in for number of daily steps via online survey form.
  Arms: Telemedicine
Behavioral: Lifestyle — All participants will be educated on physical activity recommendations, including achieving a minimum of 12,000 steps daily, and required to perform weekly check-in for number of daily steps via online survey form.
  Arms: Lifestyle

SUMMARY:
The goal of this clinical trial is to learn if telemedicine exercise programme can improve the cardiorespiratory fitness (how well your body delivers oxygen to muscles and organs) and insulin resistance in Asian children with low cardiorespiratory fitness levels. The main questions it aims to answers are:

* Does telemedicine exercise programme improve the number of 20-metre laps the participant is able to run?
* Does telemedicine exercise programme improve the insulin sensitivity using the Homeostatic Model Assessment for Insulin Resistance (HOMA-IR) formula?

Researchers will compare the telemedicine exercise programme to current active lifestyle programme (e.g., daily step count monitoring) to see if telemedicine exercise programme is more effective in improving cardiorespiratory fitness.

Participants will:

* participate in weekly telemedicine exercise programme or adhere to current active lifestyle recommendations through daily step count reporting for 10 weeks
* visit the clinic for pre- and post-programme cardiorespiratory fitness assessments and blood taking

DETAILED DESCRIPTION:
This study is to investigate the effectiveness of delivering exercise intervention programme to improve cardiorespiratory fitness through telemedicine for paediatric patients with low cardiorespiratory fitness levels. Conventionally, exercise programme for these patients are conducted within hospital premises. However, some challenges may deter patients from enrolling into these programmes, such as long travelling distance, lack of available caregiver and unsuitable timings. Understanding the impact of a shorter-term programme (i.e., 10-week programme) on cardiorespiratory fitness and glucose metabolism also allows us to customise programmes of appropriate length to deliver the require health impact instead of subjecting all patients to a lengthy programme. Therefore, evaluating the effectiveness of telemedicine-based exercise programme will enable us to fine-tune our programme and provide an alternative mode of exercise intervention so as to cater for a wider range of paediatric patients.

ELIGIBILITY:
Inclusion Criteria:

* 12 to 17 years (secondary school students)
* able to participate in school physical education lessons

Exclusion Criteria:

* less than 12 years or older than 17 years (non-secondary school students)
* has medical or musculoskeletal condition(s) preventing participation in school physical education lessons or exercise

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 122 (Estimated)
Dates: Start 2025-05-02 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Cardiorespiratory fitness assessment | At the end of 10-week programme
  Cardiorespiratory fitness (CRF) is defined by the number of completed laps in Progressive Aerobic Cardiovascular Endurance Run (PACER) test, corresponding to the respective CRF levels for gender

SECONDARY OUTCOMES:
Insulin resistance | At the end of the 10-week programme
  Insulin sensitivity is defined by the HOMA-IR formula [(fasting insulin in µU/ml) x (fasting glucose in mmol/L) / 22.5]; normal is < 2.5

CONTACTS AND LOCATIONS:
Overall Officials: Benny Loo, Principal Investigator — KK Women's and Children's Hospital
Locations (1):
- KK Women's and Children's Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No
The data generated and/or analysed during this study are not publicly available due to institutional policy on data confidentiality but are available from the corresponding author on reasonable request.

REFERENCES:
- [Background] Hall LM, Moran CN, Milne GR, Wilson J, MacFarlane NG, Forouhi NG, Hariharan N, Salt IP, Sattar N, Gill JM. Fat oxidation, fitness and skeletal muscle expression of oxidative/lipid metabolism genes in South Asians: implications for insulin resistance? PLoS One. 2010 Dec 1;5(12):e14197. doi: 10.1371/journal.pone.0014197. PMID 21152018
- [Background] Fedewa MV, Gist NH, Evans EM, Dishman RK. Exercise and insulin resistance in youth: a meta-analysis. Pediatrics. 2014 Jan;133(1):e163-74. doi: 10.1542/peds.2013-2718. Epub 2013 Dec 2. PMID 24298011
- [Background] Berman LJ, Weigensberg MJ, Spruijt-Metz D. Physical activity is related to insulin sensitivity in children and adolescents, independent of adiposity: a review of the literature. Diabetes Metab Res Rev. 2012 Jul;28(5):395-408. doi: 10.1002/dmrr.2292. Epub 2012 Mar 2. PMID 22389103
- [Background] Schmitz KH, Jacobs DR Jr, Hong CP, Steinberger J, Moran A, Sinaiko AR. Association of physical activity with insulin sensitivity in children. Int J Obes Relat Metab Disord. 2002 Oct;26(10):1310-6. doi: 10.1038/sj.ijo.0802137. PMID 12355326
- [Background] Ruiz JR, Cavero-Redondo I, Ortega FB, Welk GJ, Andersen LB, Martinez-Vizcaino V. Cardiorespiratory fitness cut points to avoid cardiovascular disease risk in children and adolescents; what level of fitness should raise a red flag? A systematic review and meta-analysis. Br J Sports Med. 2016 Dec;50(23):1451-1458. doi: 10.1136/bjsports-2015-095903. Epub 2016 Sep 26. PMID 27670254
- [Background] Wong PC, Chia MY, Tsou IY, Wansaicheong GK, Tan B, Wang JC, Tan J, Kim CG, Boh G, Lim D. Effects of a 12-week exercise training programme on aerobic fitness, body composition, blood lipids and C-reactive protein in adolescents with obesity. Ann Acad Med Singap. 2008 Apr;37(4):286-93. PMID 18461212
- [Background] Santos R, Mota J, Okely AD, Pratt M, Moreira C, Coelho-e-Silva MJ, Vale S, Sardinha LB. The independent associations of sedentary behaviour and physical activity on cardiorespiratory fitness. Br J Sports Med. 2014 Oct;48(20):1508-12. doi: 10.1136/bjsports-2012-091610. Epub 2013 Feb 14. PMID 23410883
- [Background] Calcaterra V, Verduci E, Vandoni M, Rossi V, Di Profio E, Carnevale Pellino V, Tranfaglia V, Pascuzzi MC, Borsani B, Bosetti A, Zuccotti G. Telehealth: A Useful Tool for the Management of Nutrition and Exercise Programs in Pediatric Obesity in the COVID-19 Era. Nutrients. 2021 Oct 20;13(11):3689. doi: 10.3390/nu13113689. PMID 34835945
- [Background] Takken T, Bongers BC, van Brussel M, Haapala EA, Hulzebos EHJ. Cardiopulmonary Exercise Testing in Pediatrics. Ann Am Thorac Soc. 2017 Jul;14(Supplement_1):S123-S128. doi: 10.1513/AnnalsATS.201611-912FR. PMID 28398090
- [Background] Tomkinson GR, Lang JJ, Tremblay MS, Dale M, LeBlanc AG, Belanger K, Ortega FB, Leger L. International normative 20 m shuttle run values from 1 142 026 children and youth representing 50 countries. Br J Sports Med. 2017 Nov;51(21):1545-1554. doi: 10.1136/bjsports-2016-095987. Epub 2016 May 20. PMID 27208067
- [Background] Tomkinson GR, Lang JJ, Blanchard J, Leger LA, Tremblay MS. The 20-m Shuttle Run: Assessment and Interpretation of Data in Relation to Youth Aerobic Fitness and Health. Pediatr Exerc Sci. 2019 May 1;31(2):152-163. doi: 10.1123/pes.2018-0179. Epub 2019 Mar 18. PMID 30885058
- [Background] Hui SS, Zhang R, Suzuki K, Naito H, Balasekaran G, Song JK, Park SY, Liou YM, Lu D, Poh BK, Kijboonchoo K, Thasanasuwan W. Physical activity and health-related fitness in Asian adolescents: The Asia-fit study. J Sports Sci. 2020 Feb;38(3):273-279. doi: 10.1080/02640414.2019.1695334. Epub 2019 Nov 27. PMID 31774367
- [Background] Hogstrom G, Nordstrom A, Nordstrom P. High aerobic fitness in late adolescence is associated with a reduced risk of myocardial infarction later in life: a nationwide cohort study in men. Eur Heart J. 2014 Nov 21;35(44):3133-40. doi: 10.1093/eurheartj/eht527. Epub 2014 Jan 7. PMID 24398666
- [Background] Ruiz JR, Castro-Pinero J, Artero EG, Ortega FB, Sjostrom M, Suni J, Castillo MJ. Predictive validity of health-related fitness in youth: a systematic review. Br J Sports Med. 2009 Dec;43(12):909-23. doi: 10.1136/bjsm.2008.056499. Epub 2009 Jan 21. PMID 19158130
- [Background] Ortega FB, Ruiz JR, Castillo MJ, Sjostrom M. Physical fitness in childhood and adolescence: a powerful marker of health. Int J Obes (Lond). 2008 Jan;32(1):1-11. doi: 10.1038/sj.ijo.0803774. Epub 2007 Dec 4. PMID 18043605
- [Background] Raghuveer G, Hartz J, Lubans DR, Takken T, Wiltz JL, Mietus-Snyder M, Perak AM, Baker-Smith C, Pietris N, Edwards NM; American Heart Association Young Hearts Athero, Hypertension and Obesity in the Young Committee of the Council on Lifelong Congenital Heart Disease and Heart Health in the Young. Cardiorespiratory Fitness in Youth: An Important Marker of Health: A Scientific Statement From the American Heart Association. Circulation. 2020 Aug 18;142(7):e101-e118. doi: 10.1161/CIR.0000000000000866. Epub 2020 Jul 20. PMID 32686505